CLINICAL TRIAL: NCT03599167
Title: Evaluation of the Compliance to HAS 2014 (Haute Autorité de Santé) Guidelines for Red Blood Cells Transfusion in Preterm Infant in a French Neonatal Intensive Care Unit
Brief Title: Red Blood Cell Transfusion in Very Premature Infants and HAS 2014 Guideline
Acronym: RBCPREM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI01-MME-BESSARION
Record Dates: First submitted 2018-07-05; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Practice Guideline of Erythrocyte Transfusion in Preterm Infant
Keywords: red blood cell transfusion; preterm infant; HAS guideline; transfusion guidelines; kappa agreement test application
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The indications that motivated the decision to transfuse (or not) were analyzed to verify compliance with HAS recommendations. Medical records from 57 premature infants < 32 weeks hospitalized between 2016 -2017 were retrospectively analysed, especially all the events related to monitoring of hemoglobin level and RBC transfusions during the first month of life. The criteria (postnatal age, rate of haemoglobin, type of breathing assistance, oxygen needing, medullary regeneration) on which rely the decision process in the HAS algorithm for the RBC transfusion were also considered, as well as the final decision actually adopted for each case (transfused/ not transfused). All this made it possible to determine the kappa coefficient for evaluation of agreement with HAS new guidelines in the investigator's medical staff.

ELIGIBILITY:
Inclusion Criteria:

* preterm infant hospitalized in Amiens School hospital (CHU Amiens-Picardie) between October 2016 and April 2017 during the first month of life, with allowed access on data recorded in medical files concerning the evolution of clinical characteristics (body weight,…) and the results of laboratory analyses performed during this initial hospital stay.

Exclusion Criteria:

* less than 25 weeks or more than 32 weeks at birth
* any hemoglobin dosage during the hospital stay
* serious congenital malformation
* known or documented neonatal red blood cell disease (inherited hemolysis, enzymopathy of red blood cell membrane,…)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: preterm infant hospitalized in Amiens School hospital (CHU Amiens-Picardie) between October 2016 and April 2017 during the first month of life
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Proportion of events managed in accordance with the HAS guidelines for RBC tranfusion in the very preterm infants (< 32 weeks). | during the first month of life

SECONDARY OUTCOMES:
Evolution of the haemoglobin level (Hematocrit) | during the first month of life
  from the birth until the day 28, with respect to postnatal age and the gestational age
volume of blood loss | during the first month of life
number of transfusion during the first month of life | during the first month of life
correlation between the number of transfusion and the volume of blood loss | during the first month of life
Analyses of neonatal morbidity associated with blood transfusion in premature neonates under 32 weeks of pregnancy | during the first month of life
  Neonatal morbidity are patent ductus arterious, intraventricular hemorrhage, chronic lung disease, necrotizing enterocolitis, retinopathy of the prematurity, materno-fetal infection and the late-onset infection, and diverse hematological practices

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France